CLINICAL TRIAL: NCT03641417
Title: BARI-INSIGHT: A Double-blind, Placebo-controlled, Within-subject, Cross-over Mechanistic Study Investigating the Role of Ghrelin in Regulating Appetite and Energy Intake in Patients Following Bariatric Surgery
Brief Title: Investigating the Role of Ghrelin in Regulating Appetite and Energy Intake in Patients Following Bariatric Surgery (BARI-INSIGHT)
Acronym: BARI-INSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17/0887
Record Dates: First submitted 2018-08-01; First posted 2018-08-22 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Bariatric Surgery Candidate; Appetitive Behavior
Keywords: Obesity; Bariatric surgery; Appetite; Ghrelin; Energy intake; Gut hormones; Adipokines
MeSH Terms: conditions — Obesity; Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled, within-subject, crossover mechanistic study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLWL-01 (Experimental): Oral administration of GLWL-01 300mg BD for 10 days
  Interventions: Drug: GLWL-01
- Placebo (Placebo Comparator): Identical oral capsules with no active ingredient, administered BD for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GLWL-01 — Small molecule inhibitor of Ghrelin-O-Acyltransferase (GOAT) to reduce levels of circulating acyl ghrelin.
  (Defined as a mechanistic study by MHRA; intervention not for therapeutic purposes in this study.)
  Arms: GLWL-01
Other: Placebo — Same as GLWL-01, but no active ingredient
  Arms: Placebo

SUMMARY:
Bariatric surgery helps patients with severe obesity to lose weight, cures and prevents diseases linked to obesity and reduces the risk of death. Unfortunately, 1 in 5 patients do not respond well to surgery in terms of weight loss and health gains. Thus, maximising weight loss and health benefits after surgery is critical. This study aims to gain insight into the role that the appetite-stimulating hormone, ghrelin, plays in driving appetite and energy intake in patients with poor weight loss (≤ 20% total body weight) following bariatric surgery. This will guide future work to develop pharmacological treatments for obesity, both as standalone treatments and adjuncts to bariatric surgery.

Participants will be invited to attend the Clinical Research Facility at University College London Hospital for a screening visit and six study visits. Active ghrelin levels will be reduced by inhibiting ghrelin-o-acyl-transferase (GOAT), the enzyme needed to generate active ghrelin (acyl ghrelin, AG). Participants will be randomised to receive GLWL-01 (GOAT inhibitor) 300mg BD or placebo for a 10 day study cycle. The effect of AG reduction on appetite and energy intake will be evaluated through both fixed-energy and ad libitum meal tests on day 7 and 10, respectively. Measures of body weight and composition, appetite and food cravings will be performed in addition to biochemical profiling of circulating gut hormone, adipokine and cytokine levels. Targeted physical examinations and assessment of adverse events will be performed. Safety monitoring calls will be conducted 2 and 7 days after the last dose. Following a 6-10 week washout period, participants will cross over to receive either placebo or GLWL-01 300mg BD and undergo a second study cycle, with all measures repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 64 years inclusive.
2. Minimum 1 year since primary RYGB or primary SG.
3. Poor weight-loss (≤20% total body WL) not attributable to a surgical or psychological cause.
4. Suboptimal nutrient-stimulated AG level assessed by a screening meal test. Suboptimal ghrelin response is defined as AG:DAG ratio (expressed as a percentage) of >10% and/or failure to suppress AG (i.e. <20%) in response to a standard 500kcal liquid meal.
5. Weight-stable for at least 3 months prior to screening, determined by ≤5 % variation in body weight over this time.
6. BMI ≤60 kg/m2
7. Females of childbearing potential and males must be willing to use highly effective methods of contraception, with two methods preferred, from the time consent is signed until 8 weeks after treatment discontinuation (Appendix 2).
8. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for trial treatment. NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
9. Able to read and write in English.
10. Willing and able to provide written informed consent and comply with the study protocol.

Exclusion Criteria:

1. Had a primary bariatric surgery procedure other than gastric bypass and sleeve gastrectomy, or revisional bariatric surgery of any operation type.
2. Participation in other clinical intervention trial at any time during recruitment and study execution.
3. Participation in a clinical trial within 30 days (defined as last dose of study drug) prior to GLWL-01 first dose.
4. Eli Lilly and Company or GLWL Research Inc. employees, investigators or site personnel directly affiliated with this study, and their immediate family. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
5. Weight exceeding 200kg (due to limitations of body composition analyser employed in the BARI-OPTIMISE Trial)
6. Pregnant or lactating mothers.
7. Known or suspected hypersensitivity to GLWL-01 450mg 300mg and placebo or any of the excipients involved in their formulation.
8. Active diabetes mellitus, type 1 or 2

   a) Patients with complete remission of diabetes are however eligible. Complete remission is defined as return to normal measures of glucose metabolism (HbA1c <6.5%, fasting glucose <5.6 mmol/l) of at least 1 year's duration in the absence of active pharmacological therapy or ongoing procedures.
9. History of clinically overt uncontrolled or untreated endocrine illness such as pituitary, adrenal or thyroid disease.
10. Clinically significant cardiovascular abnormality:

    1. Unstable hypertension, clinically significant ECG abnormalities, liver cirrhosis.
    2. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
    3. Known cardiac arrhythmia, including if asymptomatic or previous history of arrhythmia.
    4. Heart rate ≥ 100 beats/minute at screening on two separate measurements.
    5. History of stroke, unstable angina, acute coronary syndrome, congestive heart failure New York Heart Association class III-IV within the preceding 12 months.
    6. Have an abnormality in the 12-lead ECG, including corrected QT interval with Frederica's correction (QTcF) >450 msec for men and >470 msec for women or an abnormality that, in the opinion of the investigator, increases the risks associated with participating in the study. If QTcF does not meet criteria, ECGs may be repeated once after 5 minutes of rest.
11. Renal impairment (estimated glomerular infiltration rate eGFR <60 ml/min 1.73 m2)
12. History or evidence of liver disease

    1. Chronic disease: including but not limited to chronic alcoholic liver disease, cirrhosis of any cause or chronic autoimmune hepatitis.
    2. Acute disease: recent history (within 3 months of screening) of acute viral hepatitis
    3. Liver function test values (AST, ALT, GGT, ALP) > 3x the upper normal limit
13. History of biliary disease including primary sclerosing cholangitis.

    a) Patients with a history of cholecystectomy more than 6 months prior to screening are eligible for recruitment.
14. History of pancreatitis.
15. Evidence of human immunodeficiency virus (HIV) infection, hepatitis B, hepatitis C and/or positive results at screening for the respective antibodies for HIV, hepatitis B surface antigen, or hepatitis C antibodies.
16. Evidence of significant active or unstable/uncontrolled psychiatric disease by medical history.

    1. Lifetime history of suicidal behaviour or severe depression assessed by direct questioning and review of medical history.
    2. Patients whose disease state is considered stable and expected to remain stable throughout the course of the study, in the opinion of the investigator, may be considered for inclusion if they are not on excluded medications.
17. Use of weight loss medications within 30 days of first dose of study medication.
18. Concomitant usage of GLP-1 receptor agonist/DPPIV-inhibitors/insulin.
19. Unable to refrain from or anticipates the use of:

    1. Any drugs known to be significant inhibitors of cytochrome P450 (CYP)3A enzymes and/or P-glycoprotein (P-gp) including regular consumption of grapefruit or grapefruit juice for 14 days prior to the first dose of study medication and throughout the study. Appropriate sources will be consulted by the principal investigator (PI) or designee to confirm lack of pharmacokinetic (PK) or pharmacodynamic (PD) interaction with study medication. Paracetamol (up to 2 grams per 24-hour period) may be permitted during the study.
    2. Any drugs known to be significant inducers of CYP3A enzymes and/or P-gp, including St. John's Wort, for 28 days prior to the first dose of study medication and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/PD interaction with study medication.
20. Currently taking simvastatin >10 mg per day, atorvastatin >20 mg per day, or lovastatin >20 mg per day. The doses of these statins in combination products should not exceed these defined dose levels. Patients with a history of statin-induced myopathy/rhabdomyolysis should also be excluded.
21. Regular user of known drugs of abuse and/or shows positive findings on urinary drug screening.
22. An average weekly alcohol intake that exceeds 21 units per week (males ≤65 years of age) and 14 units per week (females and males >65 years of age), or is unwilling to stop alcohol consumption for the duration of the study (1 unit = 360 mL of beer; 150 mL of wine; 45 mL of distilled spirits).
23. Venous access insufficient to allow for blood sampling as per the protocol.
24. Any major surgery within 60 days prior to the first dose or has planned elective surgeries to occur during the study.
25. Unsuitable for inclusion in the study in the opinion of the investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Within-subject acute energy intake | Final day of each study cycle, Day 10
  Evaluate the effect of reduced circulating AG on within-subject acute energy intake assessed during an ad libitum meal.

SECONDARY OUTCOMES:
Fasted appetite scores | Day 7 of each study cycle
  in response to a fixed meal assessed using visual analogue scales (VAS).
Area-under-the-curve for appetite scores | Day 7 of each study cycle
  in response to a fixed meal assessed using visual analogue scales (VAS).
Macronutrient selection | Daily during each study cycle
  assessed using a 24-hour diet diary and food selection during the ad libitum meal.
Subjective aspects of appetite | Final day of each study cycle, Day 10
  specifically hunger, fullness, pleasantness to eat and nausea. Assessed using VAS and food craving questionnaires.
24-hour energy intake | Final day of each study cycle, Day 10
  assessed using a 24-hour diet diary, completed daily during GLWL-01 and placebo study arms.
Gut hormones levels | Day 7 of each study cycle
  Circulating levels of gut hormones in response to a fixed meal.
Adipokine levels | Day 7 of each study cycle
  Circulating levels of adipokines in response to a fixed meal
Body weight | Final day of each study cycle, Day 10
  assessed using a bioelectrical impedance analyser (BIA).
Body composition | Final day of each study cycle, Day 10
  assessed using a bioelectrical impedance analyser (BIA).
Inflammatory markers and cytokines | Final day of each study cycle, Day 10
  Evaluate the effect of reduced circulating AG on circulating inflammatory markers and cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Batterham, PhD FRCP, Principal Investigator — UCL
Locations (1):
- University College London, London, United Kingdom